CLINICAL TRIAL: NCT06431841
Title: Postmarketing Parallel Randomized Clinical Trial to Determine the Efficacy and Safety of Atropine and DIMS Lenses in the Control of Myopia in a Pediatric Population.
Brief Title: Atropine and Spectacle Combination Treatment (ASPECT): 12-month Results of a Randomized Clinical Trial for Myopia Control
Acronym: ASPECT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Noemi Guemes, Principal Investigator and sponsor, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/522-EC_M
Record Dates: First submitted 2024-03-13; First posted 2024-05-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIMS Lenses (Experimental): Atropine 0,025% + DIMS Lenses
  Interventions: Drug: Atropine 0,025%; Device: DIMS Lenses
- Monofocal Lenses (Active Comparator): Atropine 0,025% + monofocal (single vision) Lenses
  Interventions: Drug: Atropine 0,025%; Device: Monofocal lenses

INTERVENTIONS:
Drug: Atropine 0,025% — Atropine 0,025% (1 drop per day)
Device: DIMS Lenses — Use of peripheral defocus lenses with DIMS technology, the design of which simultaneously introduces myopic defocus and provides clear vision to the wearer at all viewing distances.
  Arms: DIMS Lenses
Device: Monofocal lenses — Use of monofocal lenses.
  Arms: Monofocal Lenses

SUMMARY:
Phase IV clinical trial to evaluate whether there is a significant difference in the control of myopia progression in myopic children treated with 0.025% atropine and DIMS spectacle lenses compared to 0.025% atropine and single vision (SV) lenses. Open-label, randomized, parallel clinical trial with 2 arms, involving 111 patients in total. The primary efficacy endpoint will be the change in cycloplegic spherical equivalent refraction (SER) and axial length (AL) compared to baseline values.

ELIGIBILITY:
Inclusion criteria

* Age between 4-16 years.
* Signing of informed consent.
* Refractive error: myopia greater than -1.00 diopters (D).
* Myopia progression of at least -0.50 D in the last 12 months.
* Astigmatism of 2 D or less and anisometropia of 1.50 D or less.
* Best-corrected monocular visual acuity (VA) of 0.2 logMAR(6/9) or better.

Exclusion criteria

* Children under 4 years old and over 16 years old
* Strabismus and binocular vision anomalies.
* Alterations in eye fundus that the researcher consider necessary the patient exclution.
* Ocular pathology of the anterior segment (media opacity such as cataracts, glaucoma, aphakia, pseudophakia, uveitis, keratoconus or surface alterations), and any pathology of the posterior segment that prevents correct vision
* Amblyopia
* Previous eye surgery
* Systemic pathology (cardiopulmonary pathology, connective tissue alterations, neurological or psychiatric pathology) or baseline situation of the patient that does not allow the examination to be carried out (such as mental or psychomotor retardation)
* Previous myopia control treatments including orthokeratology, rigid contact lenses, bifocal or myopia control soft contact lenses, bifocal and multifocal ophthalmic lenses within 3 months prior to the study.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic spherical equivalent refraction (SER) change | 2 years (24 months)
  Cycloplegic spherical equivalent refraction (SER) change
Axial length (AL) change | 2 years (24 months)
  Axial length (AL) change

CONTACTS AND LOCATIONS:
Locations (1):
- Noemi Guemes, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No